CLINICAL TRIAL: NCT05910294
Title: Randomized Pilot Prevention Trial to Improve Sexual and Vulvovaginal Health Concerns in Premenopausal Female Breast Cancer Patients Receiving Ovarian Suppression
Brief Title: A Study to Prevent and Improve Sexual Health Concerns for People With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-109
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Improve Sexual Health; Improve Vulvovaginal Health
Keywords: Sexual Health Concerns; Prevention; Premenopausal; Female Breast Cancer Patients; Receiving Ovarian Suppression; 23-109
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- symptom onset (Active Comparator): Symptom onset arm will receive treatment at the time symptoms develop. Patients will be provided a list of recommended moisturizers by the female sexual medicine and women's health program (FSMWHP), but will purchase the moisturizers themselves at their local pharmacy.
  Interventions: Other: questionnaires; Other: moisturizers
- intervention (Experimental): Patients who are randomized to the upfront arm will receive sexual health counseling and be initiated on non-hormonal moisturizers 3-5 times per week (based on data regarding need in our patient population) at the time ovarian suppression. The upfront intervention group will also be educated about dilators and have a consultation with a pelvic floor physical therapist. Some potential vaginal moisturizers include Hyalogyn, Replens, Liquibeads, or Vitamin E capsules.
  Interventions: Other: questionnaires; Other: moisturizers

INTERVENTIONS:
Other: questionnaires — Vaginal Assessment Scale (VAS) & Vulvar Assessment Scale (VuAS) Breast Clinical Care and Symptom Survey (BCCSS) Female Sexual Function Index (FSFI) Sexual Activity Questionnaire (SAQ) Female Sexual Distress Scale Revised (FSDS-R) Menopausal Symptom Check List (MSCL) Patient-reported Outcomes Measurement Information System Sexual Function Instrument (PROMIS-SF) Weekly Non-Hormonal Moisturizer Diary
Other: moisturizers — Patients will be provided a list of recommended moisturizers by the female sexual medicine and women's health program (FSMWHP), but will purchase the moisturizers themselves at their local pharmacy.
  Arms: symptom onset
Other: moisturizers — potential vaginal moisturizers include Hyalogyn, Replens, Liquibeads, or Vitamin E capsules
  Arms: intervention

SUMMARY:
Researchers are doing this study to look at whether sexual health counselling and using non-hormonal moisturizer at the start of ovarian suppression may be able to prevent or reduce side effects such as vaginal dryness and sexual dysfunction. Researchers will compare how effective this prevention intervention works compared to the usual approach, which is to treat these side effects after they start. All participants will also complete surveys about their sexual health. This information will help researchers learn more about the sexual health of women with breast cancer receiving ovarian suppression.

DETAILED DESCRIPTION:
50 premenopausal or perimenopausal women who are receiving ovarian suppression as part of their breast cancer treatment will be randomized to upfront intervention vs at the time of symptom development (standard of care). Patients will have subjective and objective monitoring of vaginal dryness and sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 years of age or older
* Breast cancer patients with hormone receptor positive breast cancer , stage 0-III
* Premenopausal or perimenopausal women who have either been pregnant or had at least one menstrual period in the last 24 months or have/had an IUD in place
* Patients currently on or are being initiated on ovarian suppression
* Patients are asymptomatic for vaginal symptoms of estrogen deprivation (i.e. vaginal dryness, dyspareunia, or discomfort [pain with intercourse or examination]) and score a 3 or less on the VAS and VuAS

Exclusion Criteria:

* Postmenopausal women who have been without a period for ≥ 2 years
* Patients who score a 4 or above on the VAS and VuAS
* Patients already using VVA treatment (e.g. intravaginal estrogen, other non-hormonal moisturizer or suppository), unless discontinued with washout of 4 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a score of 4 or greater in VAS | 1 year
  measured by the Vaginal Assessment Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Shari Goldfarb, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center - Suffolk (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm